CLINICAL TRIAL: NCT05045560
Title: Study of Antenatal and Postnatal Data of Anorectal Malformations Diagnosed at Montpellier University Hospital Over a 10-year Period (2010-2020) : Why and How to Improve Antenatal Counseling ?
Brief Title: Study of Antenatal and Postnatal Data of Anorectal Malformations Diagnosed at Montpellier University Hospital Over a 10-year Period (2010-2020)
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0616
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Anorectal Malformations
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- antenatal diagnosis of anorectal malformation: Groupe 1 : antenatal diagnosis of anorectal malformation
- postnatal diagnosis of anorectal malfiormation with associated anomalies on antenatal ultrasound: Groupe 2 : postnatal diagnosis of anorectal malfiormation with associated anomalies on antenatal ultrasound
- postnatal diagnosis of anorectal malformation with anormal antenatal ultrasound: Groupe 3 : postnatal diagnosis of anorectal malformation with anormal antenatal ultrasound

SUMMARY:
Objective :

Anorectal malformations (ARMs) are part of a spectrum of malformations due to an abnormal separation between the urogenital and digestive tracts during embryonic life. The prevalence of ARM is 1/2000 - 1/5000 live births, making it a relatively common malformation.

The impact of an ARM depends mainly on the type of malformation, which can be difficult to evaluate in the antenatal period, and whether it is isolated or associated (50-80%) with other malformations or genetic syndromes. Only 1 to 16% of ARMs are diagnosed in the antenatal period.

The objective of this study is to compare cases of prenatal diagnosis of ARM, cases of postnatal diagnosis of ARM with other antenatal ultrasound abnormalities, and those with normal antenatal ultrasound, in terms of management and functional prognosis, to identify ways to improve prenatal counseling.

Materials and methods :

In this retrospective monocentric study, the investigators have included all fetuses and newborns born between January 2010 and September 2020 with anorectal malformations, diagnosed from postnatal radiological examinations and surgical or autopsy reports at the University Hospital of Montpellier. The Krickenbeck classification was used to classify the ARMs and to assess the functional prognosis.

ELIGIBILITY:
Inclusion criteria:

* fetuses and newborns born between January 2010 and September 2020 with anorectal malformations
* diagnosed from postnatal radiological examinations and surgical or autopsy reports at the University Hospital of Montpellier.

Exclusion criteria:

* foreign-born patient
* anorectal malformation associated with an abdominal wall defect

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all fetuses and newborns born between January 2010 and September 2020 with anorectal malformations, diagnosed from postnatal radiological examinations and surgical or autopsy reports at the University Hospital of Montpellier.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Number of ante or post-natal diagnosispremolars | 1 day
  Number of ante or post-natal diagnosis

SECONDARY OUTCOMES:
Number of with or without associated antenatal anomalies | 1 day
  Number of with or without associated antenatal anomalies

CONTACTS AND LOCATIONS:
Overall Officials: Florent Fuchs, MD; PHD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC